CLINICAL TRIAL: NCT00006316
Title: Discontinuation of Antifungal Therapy for Histoplasmosis Following Immunologic Response to Antiretroviral Therapy
Brief Title: Withdrawal of Antifungal Treatment for Histoplasmosis in Patients After Improved Immune Response to Anti-HIV Drugs
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: ACTG A5038; AACTG A5038
Record Dates: First submitted 2000-09-28; First posted 2001-08-31 (Estimated); Last update posted 2008-08-01 (Estimated); Status verified 2004-02

CONDITIONS: HIV Infections; Histoplasmosis
Keywords: AIDS-Related Opportunistic Infections; Histoplasmosis; Antifungal Agents; Recurrence; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections; Histoplasmosis; AIDS-Related Opportunistic Infections; Recurrence

SUMMARY:
The purpose of this study is to determine whether stopping preventive histoplasmosis medications in patients who are currently receiving effective anti-HIV drugs will place them at risk for getting histoplasmosis again.

Histoplasmosis is a serious opportunistic (AIDS-related) infection that responds well to antifungal medications. Before anti-HIV drugs, patients with histoplasmosis required lifelong antifungal therapy. Patients who take anti-HIV drugs for a long time may see an improvement in their immune system functions. Improved immune function may eliminate the need for long-term preventive treatment with antifungal agents. Doctors want to see if the improved immune functions allow preventive treatment for histoplasmosis to be stopped. (This study has been changed to include histoplasmosis treatment with drugs other than itraconazole.)

DETAILED DESCRIPTION:
Histoplasmosis is a serious opportunistic infection in persons with AIDS that demonstrates an excellent response to antifungal therapy. However, until the advent of highly active antiretroviral therapy (HAART), patients with histoplasmosis required lifelong suppressive antifungal therapy. It is thought that immune reconstitution as a result of HAART may diminish the need for chronic therapy. Histoplasmosis offers an opportunity to examine the concept of discontinuation of maintenance therapy as it is rapidly diagnosed and effectively treated with itraconazole [AS PER AMENDMENT 9/27/00: or other appropriate therapy for disseminated histoplasmosis] should relapse occur.

Patients discontinue antifungal maintenance therapy. Patients are seen for routine visits every 8 weeks and urine and serum specimens are collected for real time Histoplasma antigen testing and immunologic parameters. Patients with suspected recurrence, as determined by clinical or routine laboratory findings consistent with recurrent histoplasmosis, are reevaluated within 1 week of onset of these findings. Patients with suspected recurrence based on a serum or urine Histoplasma antigen rise of 2 units or more, in the absence of clinical or routine laboratory findings consistent with histoplasmosis, are reevaluated within 2 weeks. All patients with suspected recurrence have more frequent evaluations and additional laboratory tests. Those with negative studies resume bimonthly follow-up. All patients who develop proven (positive culture or positive fungal stain of tissues or body fluids) or probable relapse (clinical findings of relapse with an increase in antigen of 4.1 units or more, or no clinical findings but increases in antigen levels on repeated testing with the most recent antigen test demonstrating an increase in antigen of 4.1 units or more) or who experience persistent reduction of CD4 cell count to below 100/mm3 have antifungal induction therapy reinstituted. Patients remain on study for at least 12 months with regular follow-up/evaluations.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are 13 years or older.
* Have consent of parent or guardian if under 18 years of age.
* Have HIV infection.
* Have 2 CD4 cell counts above 150 cells/mm3 (1 of which has been obtained within 6 months and the other within 30 days before entry). Note: The 2 CD4 counts used for eligibility must be from tests performed at least 1 week apart.
* Have received at least 1 year of treatment for histoplasmosis. (This study has been changed to include patients who have received histoplasmosis treatment with drugs other than itraconazole.)
* Are receiving treatment for histoplasmosis or have stopped treatment within 24 weeks of study entry.
* Have had histoplasmosis before but are free of any signs of histoplasmosis at entry into the study.
* Have a negative pregnancy test within 14 days of study entry.
* Have been on anti-HIV drugs for at least 24 successive weeks and have been on a stable anti-HIV drug combination for at least 8 weeks before entry.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have any recurrence of histoplasmosis within 4 weeks of study entry.
* Have received medications that affect the immune system including chemotherapy or corticosteroids within the last 2 months. (This study has been changed. Patients taking IL-2 are no longer excluded.)
* Have a systemic infection. Patients on stable preventive treatment for certain opportunistic (AIDS-related) infections for at least 3 months will be eligible.
* Require treatment for fungal infections with systemic antifungal medications.
* Have meningitis or brain or spinal cord damage thought to be caused by Histoplasma infection.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50

CONTACTS AND LOCATIONS:
Overall Officials: Mitch Goldman, Study Chair; Judy Aberg, Study Chair
Locations (13):
- United States (13):
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Emory Univ, Atlanta, Georgia
  - Cook County Hosp, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana / Life Care Clinic, Indianapolis, Indiana
  - Wishard Hosp, Indianapolis, Indiana
  - Univ of Nebraska Med Ctr, Omaha, Nebraska
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Univ of Cincinnati, Cincinnati, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Texas, Southwestern Med Ctr of Dallas, Dallas, Texas